CLINICAL TRIAL: NCT02845479
Title: Pioneering Pre- and Post-Operative Integrative Care to Improve Thoracic Cancer Quality of Care: The Thoracic Peri-Operative Integrative Surgical Care Evaluation (POISE) Trial- Stage I
Brief Title: The Thoracic Peri-Operative Integrative Surgical Care Evaluation (POISE) Trial- Stage I
Acronym: POISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Ottawa Hospital Research Institute (Other); Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150449-01H
Record Dates: First submitted 2016-07-13; First posted 2016-07-27 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Lung Neoplasms; Esophageal Neoplasms; Stomach Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative Care Intervention (Experimental): Broad-based, multi-agent integrative care program delivered by naturopathic doctors (ND) in conjunction with standard surgical and oncologic care.
  Interventions: Other: Integrative Care

INTERVENTIONS:
Other: Integrative Care — Standardized supplemental/natural health product, physical, nutritional and mental/emotional recommendations based on the phases of standard care (neo-adjuvant, perioperative, adjuvant and long-term maintenance).

SUMMARY:
Stage I of the Thoracic-POISE study will pilot-test a broad-based, multi-agent integrative care intervention delivered by naturopathic doctors in conjunction with standard surgical and oncologic care of people with thoracic cancer.

DETAILED DESCRIPTION:
Despite enormous advances in thoracic surgery and oncology, two critical issues concern patients undergoing curative-intent surgery for lung, gastric and esophageal cancer: first, a majority (~60%) of patients experience minor and major adverse events occurring during and in the days following surgery; second, patients worry about the significant risk of cancer recurrence and mortality months to years after surgery. These issues, combined with side effects of chemotherapy and radiation, have detrimental effects on health-related quality of life (HRQoL). On a deeper level, there is the problem of an ongoing failure to integrate and evaluate the best of what complementary medicine has to offer surgical oncology care.

The Thoracic-POISE Project has the overarching goal of improving care for thoracic cancer patients by impacting HRQoL, reducing surgical adverse events, prolonging overall survival and pioneering integrative care delivery. This multi-stage project aims to design, pilot-test and evaluate a broad-based, multi-agent, evidence-based integrative care program to be delivered by naturopathic doctors (ND) in conjunction with standard surgical and oncologic care. It is hypothesized that this integrative care program will improve HRQoL as well as reduce surgical adverse events and improve cancer survival. Stage I of the project will pilot-test the intervention and outcomes collection in a single-arm, feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Adults eligible and scheduled for major thoracic surgery for lung, gastric or esophageal cancer
* Candidate for complete resection
* Willingness to include an integrative component to their care
* Availability for follow-up visits over the course of one year
* Willingness to be interviewed regarding their experience of care
* Ability to answer self- and interviewer- administered questions in English or French
* Understand and sign a written informed consent form in English or French

Exclusion Criteria:

* Small cell, carcinoid, or gastrointestinal stromal (GIST) tumours
* History of cancer in the last 3 years
* Already seeing a ND or involved in an integrative program of care in the last 3 months that includes complementary medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of study protocol | Enrollment - 1 year post surgery
  Percentage of participants who complete all assessments and integrative care appointments

SECONDARY OUTCOMES:
Compliance: supplemental intervention | Enrollment - 1 year post surgery
  Count of missed doses assessed by patient diary.
Compliance: nutritional intervention | Enrollment - 1 year post surgery
  Mediterranean diet score calculated by food frequency questionnaire administered at enrollment and 1 year post surgery
Compliance: physical intervention | Enrollment - 1 year post surgery
  Extent of adherence to physical activity recommendations assessed using a patient diary.
Compliance: mental/emotional domain | Enrollment - 1 year post surgery
  Number of days audio-recordings were used assessed by patient diary.
Communication between practitioners | Enrollment - 1 year post surgery
  Number of communications (phone, consult note, etc.) between integrative and standard care practitioners per participant
Qualitative experience of care and study protocol | Enrollment - 1 year post surgery
  Semi-structured interviews with thematic analysis
Feasibility of recruitment | Enrollment
  Percentage of participants recruited out of potentially eligible patients invited.

OTHER OUTCOMES:
Adverse events | Enrollment - 1 year post surgery
  Collection of adverse events related to surgery, adjuvant therapy, and the interventions
Health Related Quality of Life | Enrollment - 1 year post surgery
  Functional Assessment of Cancer Therapy-General Score
Cancer-related symptoms | Enrollment - 1 year post surgery
  Edmonton Symptom Assessment Scale
Anxiety and Depression | Enrollment - 1 year post surgery
  Hospital Anxiety and Depression Scale
Fatigue | Enrollment - 1 year post surgery
  Multidimensional Fatigue Inventory
Functional exercise capacity | Enrollment - 1 year post surgery
  6 minute walk test
Inflammation: Multi-analyte cytokine array. | Enrollment - 1 year post surgery
  Plasma concentrations of a panel of cytokines (IL2, IL10, TGF-beta, TNF-alpha, IFN-alpha, and IFN-gamma) will be measured in blood samples collected 4 weeks before surgery, 2-3 days before surgery, on post-operative day (POD) 1, POD 5 (+/-2), 3-4 weeks, 6 months and 1 year post-surgery
Natural kill cell activation | Enrollment - 1 year post surgery
  NK cell activity will be measured by NKVue™ in blood samples collected 4 weeks before surgery, 2-3 days before surgery, on post-operative day (POD) 1, POD 5 (+/-2), 3-4 weeks, 6 months and 1 year post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dugald MR Seely, ND, MSc, Principal Investigator — Canadian College of Naturopathic Medicine; Andrew JE Seely, MD, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - Ottawa General Hospital, Ottawa, Ontario
  - Ottawa Integrative Cancer Centre, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No